CLINICAL TRIAL: NCT04922333
Title: Bisphosphonate Use to Mitigate Bone Loss Secondary to Bariatric Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00074763; U01AR080969 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bone Loss
Keywords: bariatric surgery; bisphosphonate; mitigate bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and study staff will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bisphosphonate (Experimental): Participants in this arm will receive six months of 150 mg once monthly oral risedronate
  Interventions: Drug: Risedronate
- Placebo (Placebo Comparator): Participants in this arm will receive six months of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risedronate — 150mg over-encapsulated risedronate
  Other Names: Actonel; Atelvia
  Arms: Bisphosphonate
Drug: Placebo — Capsules containing placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this research study is to see whether receiving a bisphosphonate medication called risedronate can reduce bone and muscle loss following bariatric surgery. Participation will involve up to 6 study visits and last about 1 year. Risedronate is a medication that prevents bone breakdown and has been approved by the US Food and Drug Administration (FDA) for the prevention and treatment of osteoporosis in older men and women. However, risedronate has not been approved for the prevention of bone and muscle loss following vertical sleeve gastrectomy.

Participation in this study will involve completing two visits before beginning the intervention. Participants who qualify will be scheduled to begin the intervention program which will involve taking 6 monthly doses of a risedronate or placebo pill. Participants will then receive monthly contacts by study staff during this time to remind participants to take the intervention pill and ask about any adverse events. After the completion of intervention period, participants will complete up to 4 follow up study visits at 6 months (2 visits) and at 12 months (2 visits).

DETAILED DESCRIPTION:
The main objective of the proposed study is to definitively test whether risedronate use can effectively counter SG associated bone loss. To do this, we propose to randomize 120 middle-aged and older (≥40 years) SG patients to six months of risedronate or placebo treatment, with musculoskeletal outcomes assessed at baseline, six, and 12 months. Due to its robust change following SG and clinical utility in predicting fracture, our primary outcome is change in total hip areal (a)BMD measured by dual energy x-ray absorptiometry (DXA). This will be complemented by DXA-acquired aBMD assessment at other skeletal sites and appendicular lean mass, as well as quantitative computed tomography (QCT) derived changes in bone (volumetric BMD, cortical thickness, and strength) and muscle (cross sectional area, fat infiltration) at the hip and spine, and high-resolution peripheral quantitative computed tomography (HR-pQCT) derived changes in bone microarchitecture, density, and strength at the tibia and radius - allowing for novel assessment of intervention effectiveness on several state-of-the-art bioimaging metrics. Select measures of muscle function (fast 400-m walk, stair climb, knee extensor strength) are also included as proxies of fall risk. Finally, biomarkers of bone turnover (CTX, P1NP), bone-muscle crosstalk (TGF-β, RANKL, myostatin), and gut hormones (ghrelin, PYY, GLP-1) will be assessed in a tertiary aim, providing mechanistic insight into intervention-related changes to the bone-muscle unit. Thus, we aim to:

Aim 1: Determine the effect of risedronate compared to placebo on 12-month change from baseline in total hip aBMD following SG. We hypothesize that participants assigned to risedronate will better preserve total hip aBMD than participants assigned to placebo.

Aim 2: Determine the effects of risedronate compared to placebo on 12-month change from baseline in DXA-acquired aBMD at additional skeletal sites (femoral neck, lumbar spine, distal radius) and appendicular lean mass; QCT-derived measures of bone (volumetric BMD, cortical thickness, and strength) and muscle (cross sectional area, density, fat infiltration) at the hip and spine; HR-pQCT derived measures of bone microarchitecture, density, and strength at the tibia and radius; and muscle function (fast 400-m walk, stair climb, knee extensor strength) following SG. We hypothesize that participants assigned to risedronate will yield greater preservation/improvement in all secondary metrics than participants assigned to placebo.

Aim 3: Investigate the impact of treatment group assignment on biomarkers of bone turnover, bone-muscle crosstalk, and gut hormones to elucidate mechanisms underlying change in bone and muscle quantity and quality.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had sleeve gastrectomy
* Willing to provide informed consent
* Agree to all study procedures and assessments.

Exclusion Criteria:

* Weight greater than 450 lbs
* Regular use of growth hormones, oral steroids, or prescription osteoporosis medications;
* Known allergies to bisphosphonates
* Unstable gastric reflux requiring two or more additional doses per month of anti-reflux medication.
* Current participation in other research study
* Unable to provide own transportation to study visits
* Unable to position on scanner independently.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in Total Hip Areal Bone Mineral Density (aBMD) | baseline through Month 6
  Acquired through DXA scans.
Change in Total Hip Areal Bone Mineral Density (aBMD) | baseline through Month 12
  Acquired through DXA scans.

SECONDARY OUTCOMES:
Dual Energy X-Ray Absorptiometry (DXA)-acquired Femoral Neck Measurements | Baseline, Month 6, Month 12
DXA-acquired Lumbar Spine Measurements | Baseline, Month 6, Month 12
DXA-acquired Distal Radius Areal BMD Measurements | Baseline, Month 6, Month 12
DXA-acquired Appendicular Lean Mass Measurements | Baseline, Month 6, Month 12
Quantitative Computed Tomography (QCT) Acquired Compartmental Volumetric BMD (hip) Measurement | Baseline, Month 6, Month 12
QCT-acquired Compartmental Volumetric BMD (Spine) Measurement | Baseline, Month 6, Month 12
QCT-acquired Cortical Thickness (Hip) Measurement | Baseline, Month 6, Month 12
QCT-acquired Finite Element (FE) Strength (Hip) Measurement | Baseline, Month 6, Month 12
QCT-acquired Mid-Thigh Cross-Sectional Area (CSA) Measurement | Baseline, Month 6, Month 12
QCT-acquired Trunk Muscle Cross-Sectional Area (CSA) Measurement | Baseline, Month 6, Month 12
QCT-acquired Thigh Muscle Density Measurement | Baseline, Month 6, Month 12
QCT-acquired Thigh Fat Infiltration Measurement | Baseline, Month 6, Month 12
Physical Function Measurement (Fast Walk) | Baseline, Month 6, Month 12
  Fast-paced gait speed will be assessed using the fast 400 meter walk test. Participants will be asked to walk 10 laps of a 40 meter course (20 meters out and 20 meters back) as fast as possible and are given a maximum of 15 minutes to complete the test.
Physical Function Measurement (Stair Climb) | Baseline, Month 6, Month 12
  Stair climbing ability will be assessed by using the participant's fastest time achieved to climb 12 steps in two trials. Both tests are sensitive to intensive weight loss and predictive of fall risk.

OTHER OUTCOMES:
Biomarkers of Bone Turnover, Metabolism, and Bone-Muscle Crosstalk | Baseline, Month 6, Month 12
  Blood drawn for collection of biomarkers.
High Resolution peripheral Quantitative Computed Tomography (HRpQCT)-Acquired Distal Tibia Failure Load | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Bones Stiffness | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Radius Failure Load | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Radius Bone Stiffness | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Trabecular Number | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Trabecular Thickness | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Trabecular Separation | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Cortical Thickness | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Cortical Porosity | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Cortical Volumetric Bone Mineral Density | Baseline, Month 6, Month 12
HRpQCT-Acquired Distal Tibia Trabecular Volumetric Bone Mineral Density | Baseline, Month 6, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Beavers, PhD, MPH, RD, Principal Investigator — Wake Forest University Health Sciences; Jamy Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No